CLINICAL TRIAL: NCT01597063
Title: A Clinical Study to Evaluate the Relative Clinical Specificity Performance of the SEQureDx Trisomy Test in Pregnant Women at Low Risk for Fetal Chromosomal Aneuploidy
Brief Title: Clinical Evaluation of the SEQureDx Trisomy Test in Low Risk Pregnancies
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SQNM-T21-303
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Aneuploidy; Down Syndrome; Noninvasive Prenatal Screening
MeSH Terms: conditions — Aneuploidy; Down Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood specimens will be collected and processed to plasma. DNA will be extracted from the plasma.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- low risk pregnancies
  Interventions: Device: SEQureDx Trisomy Test

INTERVENTIONS:
Device: SEQureDx Trisomy Test — Plasma samples obtained from maternal blood will be tested using the SEQureDx Trisomy Test, an in vitro diagnostic test that measures circulating cell-free fetal DNA. The test detects the relative quantity of chromosome 21, which is associated with trisomy 21.

SUMMARY:
Pregnant women with low risk indicators for fetal chromosomal aneuploidy will be enrolled. Study blood will be collected in the first or second trimester at a scheduled prenatal screening visit, processed to plasma, and stored frozen until analysis. Each pregnancy will be followed until delivery and the birth outcome recorded.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy is 10-22 weeks gestation
* Between 18-34 years of age inclusive at estimated date of delivery
* No prenatal screening indicators for high risk including serum biochemical and ultrasound screening
* No personal or family history of Down syndrome
* Willing to provide written informed consent
* Willing to provide a whole blood sample
* Willing to provide access to medical records supporting fetal outcome

Exclusion Criteria:

* Fetal demise at the time of the blood draw
* Previous specimen donation under this protocol

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant with low risk for fetal chromosome 21 aneuploidy
Sampling Method: Probability Sample
Enrollment: 3333 (Actual)
Dates: Start 2012-07; Primary Completion 2014-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Estimate the false positive rate of SEQureDx Trisomy 21 Test | pregnancy outcome

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Grossu, MD, Study Director — Sequenom, Inc.
Locations (27):
- United States (27):
  - University of South Alabama, Mobile, Alabama
  - New Horizon Women's Care, Chandler, Arizona
  - Precision Trials, Phoenix, Arizona
  - Visions Clinical Research Tuscon, Tucson, Arizona
  - Descanso OBGYN, Glendale, California
  - Woodglen Medical Group, Glendora, California
  - White Memorial GYN/OB Medical Group, Los Angeles, California
  - Fair Oaks Women's Health, Pasadena, California
  - IGO Medical Group, San Diego, California
  - West Coast OBGYN, San Diego, California
  - Women's Health Care Research, San Diego, California
  - Women's Clinical Research, Vista, California
  - Hawaii Pacific Health, Honolulu, Hawaii
  - University of Iowa Health Care, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Spectrum Health - Maternal Fetal Medicine, Grand Rapids, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Virtua Health, Moorestown, New Jersey
  - Virtua Health, Mount Holly, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Saint Peter's Hospital, New Brunswick, New Jersey
  - Virtua Health, Sewell, New Jersey
  - Virtua Health, Voorhees Township, New Jersey
  - Providence Health Partners - Center for Clinical Research, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Magnolia OB/GYN Research Center- Recruiting, Myrtle Beach, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Upon analysis of collected samples and submission for publication, data will be shared as per journal requirements.

REFERENCES:
- [Background] Palomaki GE, Kloza EM, Lambert-Messerlian GM, Haddow JE, Neveux LM, Ehrich M, van den Boom D, Bombard AT, Deciu C, Grody WW, Nelson SF, Canick JA. DNA sequencing of maternal plasma to detect Down syndrome: an international clinical validation study. Genet Med. 2011 Nov;13(11):913-20. doi: 10.1097/GIM.0b013e3182368a0e. PMID 22005709
- [Background] Ehrich M, Deciu C, Zwiefelhofer T, Tynan JA, Cagasan L, Tim R, Lu V, McCullough R, McCarthy E, Nygren AO, Dean J, Tang L, Hutchison D, Lu T, Wang H, Angkachatchai V, Oeth P, Cantor CR, Bombard A, van den Boom D. Noninvasive detection of fetal trisomy 21 by sequencing of DNA in maternal blood: a study in a clinical setting. Am J Obstet Gynecol. 2011 Mar;204(3):205.e1-11. doi: 10.1016/j.ajog.2010.12.060. Epub 2011 Feb 18. PMID 21310373
- [Background] Palomaki GE, Deciu C, Kloza EM, Lambert-Messerlian GM, Haddow JE, Neveux LM, Ehrich M, van den Boom D, Bombard AT, Grody WW, Nelson SF, Canick JA. DNA sequencing of maternal plasma reliably identifies trisomy 18 and trisomy 13 as well as Down syndrome: an international collaborative study. Genet Med. 2012 Mar;14(3):296-305. doi: 10.1038/gim.2011.73. Epub 2012 Feb 2. PMID 22281937